CLINICAL TRIAL: NCT00474838
Title: The Effect of Intensive and Short-term Insulin Treatment on Long-term Pancreatic β-cell Function in Newly Diagnosed People With Type 2 Diabetes in Korea
Brief Title: Study To Evaluate Beta Cell Function and Glycemic Outcome by Intensive Insulin Therapy
Acronym: KIIT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kyunghee University Medical Center (Other)
Collaborators: Korea University Guro Hospital (Other); Hanyang University (Other); Inha University Hospital (Other); Ajou University (Other); Sanofi (Industry); East West Neo Medical Center (Other); The Catholic University of Korea (Other); Jeju National University Hospital (Other)
Responsible Party: Principal Investigator, Jeong-taek Woo, Professor, Kyunghee University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KIIT-KMC-0701
Record Dates: First submitted 2007-05-16; First posted 2007-05-17 (Estimated); Last update posted 2013-09-26 (Estimated); Status verified 2013-09

CONDITIONS: Type 2 Diabetes Mellitus; Pancreatic Beta Cell Function; Glucotoxicity
Keywords: type 2 diabetes mellitus; intensive insulin therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Hypoglycemic Agents; glimepiride; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oral AntiDiabetic Drug (Active Comparator): glimepiride and metformin and/or once daily glargine
  Interventions: Drug: Oral AntiDiabetic Drug (glimepiride and metformin)
- intensive insulin group (Experimental): insulin glargine insulin glulisine
  Interventions: Drug: intensive insulin group

INTERVENTIONS:
Drug: intensive insulin group — Once daily long acting insulin and preprandial rapid acting insulin injection
  Arms: intensive insulin group
Drug: Oral AntiDiabetic Drug (glimepiride and metformin) — glimepiride and metformin combined therapy
  Other Names: glimepiride(amaryl); metformin(diabex)
  Arms: Oral AntiDiabetic Drug

SUMMARY:
This randomized controlled prospective study aims to evaluate the efficacy of intensive insulin therapy for long term glycemic control and improvement or preservation of beta cell function in newly diagnosed type 2 diabetes patients.

DETAILED DESCRIPTION:
Type 2 diabetes is associated with beta cell dysfunction and insulin action at diagnosis of diabetes. Although the relative importance of these two alterations is controversial, growing evidence is swinging to the concept that there is no hyperglycemia without β-cell dysfunction. Also there is agreement that deterioration of glucose tolerance over time is associated with a progressive decrease of beta cell function.

Beside the role of genetic factor, the continuous decline in β-cell function is affected by glucotoxicity generated by hyperglycemia and lipotoxicity due to high fatty acid. A vicious cycle of hyperglycemia per se further impairs and may destroy β-cell. Recently, many reports have shown that early intensive glycemic control plays a role in the prevention of progressive ß-cell function and worsening of diabetes.

Some studies have shown that early intensive insulin therapy(IIT) to achieve near normoglycemia in new onset type 2 diabetes gives short term and long term improvement in glycemic control after discontinuation of insulin. It is suggested that long term glycemic control is associated with improvement of β-cell function.

In the unpublished previous pilot study, the investigators found that early intensive insulin therapy using multiple daily injection (MDI) or daily twice injection in newly diagnosed type 2 diabetes can significantly improve the beta cell function and facilitate further long term glycemic control. To establish the effectiveness of intensive insulin therapy for long term glycemic control and improvement of β-cell function, the investigators will perform a randomized controlled prospective study in newly diagnosed type 2 diabetes in Korea.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed drug naïve type 2 diabetic patient with typical diabetic symptom (polydipsia, polyuria, unexplained weight loss) within recent 1 year
* Initial HbA1c : 8.0 % ≤ HbA1c < 12.0%

Exclusion Criteria:

* Known contraindication to insulin glargine, insulin glulisine, metformin, glimepiride
* Patients with proliferative diabetic retinopathy
* Severe liver disease or AST, ALT ≥ 2.5 x ULN
* History of lactic acidosis
* Unstable or severe angina
* Congestive heart failure
* Chronic disease treated with continuous corticosteroid therapy
* Diagnosis of cancer
* Positive urine pregnancy test or plan to become pregnant during the clinical trial

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2007-04; Primary Completion 2012-08 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Long-term glycemic control | up to 2 years
Change of pancreatic beta cell function | up to 2 years

SECONDARY OUTCOMES:
Inflammatory marker and insulin sensitivity | up to 2 years
Time to reach target goal of blood glucose level | up to 2 year

CONTACTS AND LOCATIONS:
Overall Officials: Jeong-taek Woo, MD, PhD, Principal Investigator — Kyunghee University Medical Center
Locations (8):
- South Korea (8):
  - Hanyang University Medical Center, Guri-si, Gyeonggi-do
  - The Catholic University of Korea Bucheon St.Mary's Hospital, Bucheon-si
  - Inha University Hospital, Incheon
  - Jeju National University Hospital, Jeju-do
  - Kyunghee University Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
  - Kyung Hee University East Weast Neo Medicalcenter, Seoul
  - Ajou University Medical Center, Suwon